CLINICAL TRIAL: NCT04327570
Title: In-depth Characterisation of the Dynamic Host Immune Response to Coronavirus SARS-CoV-2
Brief Title: In-depth Immunological Investigation of COVID-19.
Acronym: COntAGIouS
Status: Recruiting | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Other Study IDs: COntAGIouS
Record Dates: First submitted 2020-03-26; First posted 2020-03-31 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-10

CONDITIONS: Coronavirus Infections
Keywords: COVID-19
MeSH Terms: conditions — Coronavirus Infections; COVID-19

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Biospecimen Retention: Samples With DNA — Blood, plasma, PBMC, BAL, lung tissue
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ICU-hospitalised COVID-19 patients: COVID-19 positive patients hospitalised in intensive care ('severe disease').
  Interventions: Other: Patient sampling
- ward-hospitalised COVID-19 patients: COVID-19 positive patients requiring hospitalisation,not on intensive care department ('non-severe').
  Interventions: Other: Patient sampling

INTERVENTIONS:
Other: Patient sampling — Blood draw, NP/rectal swab, bronchoscopy if clinically indicated, lung tissue if applicable

SUMMARY:
The COntAGIouS trial (COvid-19 Advanced Genetic and Immunologic Sampling; an in-depth characterization of the dynamic host immune response to coronavirus SARS-CoV-2) proposes a transdisciplinary approach to identify host factors resulting in hyper-susceptibility to SARS-CoV-2 infection, which is urgently needed for directed medical interventions.

DETAILED DESCRIPTION:
The overall aim of this prospective study is to provide an in-depth characterization of clinical and immunological features of patients hospitalized in UZ Leuven because of SARS-CoV-2 infection. For this purpose, clinical data and blood, nasopharyngeal/rectal swab, and if safe, bronchoalveolar lavage (BAL) fluid and lung tissue samples will be collected from PCR- or CT-confirmed COVID-19 patients, with varying degrees of disease severity. Assessed characteristics will be compared between severe and non-severe COVID-19 patients, and between COVID-19 positive and negative ('control') patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients >/= 18 years old AND
* Hospitalised with PCR-confirmed and/or CT-confirmed SARS-CoV-2 disease

Exclusion Criteria:

* Age < 18 years old
* No informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients (>18 years old) that are admitted to UZ Leuven from March 2020 until September 2026 with PCR-confirmed and/or CT-confirmed SARS-CoV-2 disease are eligible for inclusion.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-03-27 (Actual); Primary Completion 2026-03-30 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
Clinical Features | 6 months
  Description of clinical, laboratory and radiological features of illness and complications.
Immune host response at systemic level | 6 months
  Evaluation of dynamic host immune response at systemic level (immune signalling molecules in plasma, peripheral blood mononuclear cell isolation for advanced immunophenotyping and transcriptomics). Real-time analysis using CyTOF will be performed as screening, in combination with in-depth immunophenotyping.
Immune host response at local level | 6 months
  Evaluation of dynamic host immune response at systemic level (immune signalling molecules in plasma, peripheral blood mononuclear cell isolation for advanced immunophenotyping and transcriptomics).
Host genetic variation | 6 months
  Identification of host genetic variants that are associated with severity of disease.

SECONDARY OUTCOMES:
Comparison severe and non-severe COVID-19 hospitalised patients | 6 months
  Differences in baseline factors
Comparison severe and non-severe COVID-19 hospitalised patients | 6 months
  Differences in immune characteristics
Correlation of findings with outcome | 6 months
  Correlation of findings with outcome, aiming to identify early biomarkers of severe disease and putative targets for immunomodulatory therapy
Correlation of immune profiling - microbiome | 6 months
  Correlation of immune profiling with microbiome analysis of patients

CONTACTS AND LOCATIONS:
Overall Officials: Joost Wauters, MD PhD, Principal Investigator — UZ Leuven
Locations (1):
- UZ Leuven, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: Undecided